CLINICAL TRIAL: NCT00726011
Title: A Multicentre, Open-label, Long-term Efficacy and Safety Continuation Study of Subcutaneous Tetrodotoxin (TTX) for Moderate to Severe Cancer-related Pain
Brief Title: Tetrodotoxin Open-label Efficacy and Safety Continuation Study
Acronym: TEC-006OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC-006OL
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Pain; Cancer
Keywords: due; cancer treatment
MeSH Terms: conditions — Pain; Neoplasms | interventions — Tetrodotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tetrodotoxin (Experimental): There is only one arm; active treatment with TTX
  Interventions: Biological: Tetrodotoxin

INTERVENTIONS:
Biological: Tetrodotoxin — 30 µg twice daily for 4 days; repeated every two weeks as long as there is a meaningful analgesic response
  Other Names: TTX

SUMMARY:
Different pathophysiologic mechanisms are responsible for the development of chronic pain disorders. Pain pathways are triggered in part by ectopic discharges of voltage-sensitive sodium channels, which are in abundance in both the peripheral and the central nervous systems. Tetrodotoxin (TTX) is a selective blocker of Na+ channels and causes analgesia either by decreasing the propagation of action potentials by Na+ channels and/or by blocking of ectopic discharges associated with chronic pain. TTX is extracted from the puffer fish (fugu). Results from animal pharmacology studies revealed that TTX is a more potent analgesic than standard analgesic agents such as aspirin, morphine or meperidine.

At present, the management of severe cancer pain generally includes the use of opiates. This can often result in undesirable side effects, and treatment with this type of medication is not always effective. Because currently available pain-relieving therapy is unsatisfactory for many patients, there is a need for new therapeutic approaches for the management of moderate or severe cancer pain.

Recent studies indicate that intramuscular (into a muscle) or subcutaneous (under the skin) injections of tetrodotoxin (TTX) may reduce pain in cancer patients who did not respond to standard therapies.

The current proposed study (TEC-006OL) is designed to provide the option for all patients who participated in the TEC-006 study (both tetrodotoxin and placebo-treated) to receive or continue to receive tetrodotoxin treatment.

DETAILED DESCRIPTION:
Study Objectives: In cancer patients with moderate to severe pain who participated in the TEC-006 study:

Primary Objectives:

* To assess the long-term efficacy of subcutaneous tetrodotoxin (TTX) treatment in reducing the pain outcome and improving the quality of life (physical and emotional functioning).
* To assess the long-term safety and tolerability of subcutaneous tetrodotoxin (TTX).

Secondary Objective:

• To assess the duration of analgesia following repeated cycles of tetrodotoxin (TTX) treatment.

Overall Study Design:

This will be a multicentre, open-label, continuation trial of the efficacy and safety of tetrodotoxin in patients with inadequately controlled moderate to severe pain associated with cancer. All patients who participated in the TEC-006 study (tetrodotoxin and placebo-treated), who would like to continue with tetrodotoxin treatment and meet the inclusion/exclusion criteria, are eligible to receive the First Treatment Cycle for this continuation study.

The study will be conducted at all centres participating in the TEC-006 study. Patients may receive repeated cycles of treatment with tetrodotoxin. Each Treatment Cycle will consist of 4 days of treatment with 30 μg b.i.d. of tetrodotoxin injected subcutaneously. Each Treatment Cycle will last from the start of treatment to the end of the analgesic response. All patients completing the first Treatment Cycle in this protocol must meet the criteria of the Responder (First TEC-006OL Treatment Cycle) definition in order to be eligible for a second Treatment Cycle. Patient eligibility for all subsequent Treatment Cycles will be determined using the eligibility criteria for a Repeated Treatment Cycle.

Sample Size:

Up to 120 patients.

Investigational Product:

30ug TTX(Tetrodotoxin injectable) injected subcutaneously twice daily for 4 days.

Efficacy Variables:

Worst pain in last 24 hours, average pain in last 24 hours, and/or component-specific pain intensity in last 24 hours, ATC and breakthrough analgesic use, impact of pain on physical functioning (general activity, walking ability, or normal work), and emotional functioning (mood, relations with other people, or enjoyment of life).

Safety Variables:

Safety assessments will include adverse event reporting, vitals signs, physical and neurological examinations, 12-lead electrocardiogram, clinical laboratory tests.

Data Analysis Method:

An initial analysis of results of the TEC-006OL study will be completed in parallel with the TEC-006 study. Further periodic analyses will be completed every 6 months until the study is closed.

All efficacy and safety analyses will be performed for subjects that are dosed at least once in protocol TEC-006OL. All analyses performed will be descriptive. No statistics involving hypothesis testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

All patients who participated in the TEC-006 study (tetrodotoxin and placebo-treated) will be eligible for inclusion in this study provided they wish to continue to receive treatment and meet the inclusion and exclusion criteria.

NOTE: The blinded treatment assignment of patients in the TEC-006 will not be revealed to either the investigator or the patient. Patients will not be aware which treatment they received in the TEC-006 study. All patients will receive tetrodotoxin treatment in the TEC-006OL study.

A patient will be eligible or continue to be eligible for inclusion in this study (First Treatment Cycle and subsequent Treatment Cycles) only if all of the following criteria apply:

1. Male or female 18 years of age and over
2. In-patients or out-patients with a diagnosis of cancer
3. Patients must be experiencing somatic, visceral and/or neuropathic pain related to cancer.
4. Compliant to the requirements of the TEC-006 Protocol.
5. Inadequately controlled pain: Pain intensity described as 'moderate', 'severe' or 'excruciating', as assessed by the VRS during the screening/baseline period of the First Treatment Cycle, and a baseline pain intensity score of ≥4 as assessed by NRS (worst, average, or component-specific pain).
6. Meet the Responder or Clinical Responder definition for repeat cycle treatment (cycle #2 to cycle #4)
7. Life expectancy of > 3 months.
8. Ability to communicate well with the Investigator and to comply with the requirements of the entire study.

8. Willingness to give written informed consent (prior to any study-related procedures being performed) and to be able to adhere to the study restrictions, appointments and examination schedule.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Planned initiation of chemotherapy, radiotherapy or bisphosphonates within 30 days prior to enrolment.
2. Known renal disease.
3. If it has been more than 14 days since their TEC_006 End of Study Visit or their pain returned to baseline since their last tetrodotoxin treatment cycle (for repeat cycle).
4. Patient has previously completed 4 cycles of tetrodotoxin
5. If it has been more than 6 months since patient signed consent to participate in the TEC-006 OL study.
6. Use of anaesthetics.
7. Use of lidocaine, and other types of antiarrhythmic drugs.
8. Use of scopolamine and acetylcholinesterase-inhibiting drugs such as physostigmine.
9. History of CO2 retention, or SaO2 <80% either on room air or O2 of not greater than 2-4 L/min by nasal cannula.
10. Second or third degree heart block or prolonged QTc interval (corrected for rate) on screening ECG (confirmed > 450 msec on repeated occasion) or any other active cardiac arrhythmia or abnormality that would constitute a clinical risk.
11. Coagulation or bleeding defects if in the opinion of the Investigator this represents a risk to the subject considering the subcutaneous (s.c.) route of administration.
12. Known hypersensitivity to puffer fish, tetrodotoxin and/or its derivatives.
13. Received an investigational agent other than tetrodotoxin within 30 days prior to screening or who is scheduled to receive an investigational drug other than tetrodotoxin during the course of the study.
14. Females who are lactating or at risk of pregnancy (i.e., sexually active with fertile males and not using an adequate form of birth control).
15. Females with a positive pregnancy test at screening or on admission to study site.
16. Any other condition that, in the opinion of the investigators, is likely to interfere with the successful collection of the measures required for the study or poses a risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy: long-term efficacy of tetrodotoxin (TTX) in reducing pain and improving quality of life. Safety: long-term safety and tolerability of s.c. TTX | Repeat treatment for patients with meaningful analgesic response

SECONDARY OUTCOMES:
For each Treatment Cycle: the total number of days a subject meets the definition of pain response. | Repeat treatment for subjects with meaningful analgesic response

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Neil Hagen, MD, FRCPC, Study Chair — Tom Baker Cancer Centre
Locations (1):
- WEX Pharmaceuticals Inc., Vancouver, British Columbia, Canada